CLINICAL TRIAL: NCT00858481
Title: Efficacy and Safety of Different Strengths of Spinosad Topical Creme (0%, 0.5%, 1.0% or 2%) in Subjects With Pediculosis Capitis - a Dose Ranging Study
Brief Title: A Pilot Dose Ranging Study of Spinosad Creme Rinse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ParaPRO LLC (Industry)
Responsible Party: Dyal Garg, Ph.D., Principal Investigator, Hill Top Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPN-201-05; HTR-124235
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Pediculosis Capitis; Head Lice
Keywords: Pediculosis capitis; Head Lice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Vehicle control
  Interventions: Drug: Spinosad Creme Rinse - Vehicle Control
- 2 (Active Comparator): 0.5% Spinosad creme rinse
  Interventions: Drug: Spinosad Creme Rinse
- 3 (Active Comparator): 1.0% Spinosad Creme Rinse
  Interventions: Drug: Spinosad Creme Rinse
- 4 (Active Comparator): 2.0% Spinosad Creme Rinse
  Interventions: Drug: Spinosad Creme Rinse

INTERVENTIONS:
Drug: Spinosad Creme Rinse - Vehicle Control — One or two, 10-minute topical applications (7 days apart)
  Arms: 1
Drug: Spinosad Creme Rinse — 0.5% Spinosad Creme Rinse: one or two, 10-minute topical applications (7 days apart)
  Arms: 2
Drug: Spinosad Creme Rinse — 1.0% Spinosad Creme Rinse: one or two, 10-minute topical applications (7 days apart)
  Arms: 3
Drug: Spinosad Creme Rinse — 2.0% Spinosad Creme Rinse - one or two, 10-minute topical applications (7 days apart)
  Arms: 4

SUMMARY:
A pilot dose ranging study to evaluate the safety and efficacy of different strengths of Spinosad Creme versus a vehicle control.

DETAILED DESCRIPTION:
A Phase 2a, randomized, single investigational site, investigator/evaluator-blind, four-arm, parallel-group, vehicle-controlled, pilot study to evaluate the safety and efficacy of different strengths of Spinosad Creme rinse verses vehicle control.

ELIGIBILITY:
Inclusion Criteria:

* Active head lice infestation
* Male or female, 2 years of age or older
* Good general health
* Appropriately signed Informed Consent
* Subject agreement to not use any other form of lice treatment during the course of the study
* Subject agreement to not cut or chemically treat their hair between visits

Exclusion Criteria:

* History of irritation or sensitivity to pediculicides or hair care products
* Individuals with any visible skin/scalp condition that would interfere with the evaluation
* Individuals previously treated with a pediculicide within 4 weeks prior to study enrollment
* Individuals using hair dyes, bleaches, permanent waves or relaxing solutions 2 weeks prior to study enrollment
* Individuals who have participated in any clinical trial within 30 days of enrollment
* Individuals with family members who were infested with lice but were unwilling or unable to enroll in the study or use a standard course of lice treatment
* Females who were pregnant or nursing
* Sexually active females not using effective contraception

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of various doses of Spinosad, based on the presence or absence of live lice at 7 and 14 days post-treatment. The efficacy evaluation was performed by a trained evaluator. | 14 days

SECONDARY OUTCOMES:
Safety of various doses of Spinosad, based on the occurrence of adverse events, especially scalp irritation. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Dyal Garg, Ph.D., Principal Investigator — Hill Top Research
Locations (1):
- Hill Top Research, West Palm Beach, Florida, United States